CLINICAL TRIAL: NCT06817213
Title: Patient-Centered Decision Support for Eosinophilic Esophagitis: A Pilot Study
Brief Title: Patient-Centered Decision Support for Eosinophilic Esophagitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Joy Chang, Assistant Professor of Internal Medicine, University of Michigan
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00257119; 1K23DK129784-01A1 (NIH)
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Eosinophilic Esophagitis
Keywords: tailored educational materials; general educational materials; online surveys; decision aid
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Intervention Model Description: Participants (n-20) will be enrolled into the control arm (general education about EoE), then 20 patients will go into the DA arm. Providers will not be formally consented to have their clinics screened for participants. The study team will coordinate with Gastroenterology and Allergy providers about the initiation of the study. Providers will be informed that the study is launching and given the opportunity to "opt-out".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- General education control group (Active Comparator): General educational materials
  Interventions: Behavioral: General education control
- Decision support tool group (Experimental): Tailored educational materials
  Interventions: Behavioral: Decision support tool

INTERVENTIONS:
Behavioral: General education control — Participants will complete an online survey before reviewing education material for eosinophilic esophagitis, prior to patient's clinical physician's appointment (this appointment is a standard of care visit). Participants will complete a follow-up survey approximately 3 months after the clinic appointment.
  Arms: General education control group
Behavioral: Decision support tool — Participants will complete an online survey before reviewing tailored educational materials for eosinophilic esophagitis prior to patient's clinical physician's appointment (this appointment is a standard of care visit). The intervention is a tailored, electronic decision support intervention with a patient-facing decision aid (DA) with three components-EoE knowledge/education, values clarifications, and communication. Tailored feedback from the patient will be given to the patient's provider prior to the visit to facilitate shared decision-making in the visit. Participants will complete a follow-up survey approximately 3 months after the clinic appointment.
  Arms: Decision support tool group

SUMMARY:
The study team is conducting this project to learn more about how patients with eosinophilic esophagitis (EoE) like to use and receive educational materials about treatment options and treatment decision making.

This study will assess the efficacy of a decision support intervention to make decisions about treatment and disease management for patients with EoE and will assess the feasibility and acceptability of the intervention to inform future R01-level studies.

The study team hypothesize that deploying the intervention will be feasible, and it will demonstrate high acceptability among EoE patients. Additionally, that patients that use the intervention (vs general education about EoE) will report greater treatment knowledge, increased readiness to choose a therapy, adherence to therapy, and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* New EoE patient evaluations ≥18 years old at University of Michigan (UM) that have an upcoming outpatient visit in a UM-gastroenterology or allergy & immunology clinic,
* Able to speak and read English.

Exclusion Criteria:

* Prisoners and institutionalized individuals due to logistical limitations for use of a web app and follow-up interactions in these populations.
* Patients that have significant cognitive or visual impairment that limits interaction with the decision aid (DA)
* Patients that are terminally ill
* Patients that do not have an email address or reliable access to the internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility: measured as the proportion of eligible patients that consent to participate in the study | Recruitment period approximately 18 months
  The study aims to achieve at least 20% consented for eligible patients.
Acceptability: measured on a 4-point Likert scale | Approximately 4 months
  Measured on a 4-point Likert-scale (1) Very Unhelpful to (4) Very Helpful. Analyzed as high scores indicate more helpful.

SECONDARY OUTCOMES:
Effectiveness (within-subjects) | Day 1 up to approximately 1 month (after consent prior to standard of care clinic visit)
  Objective eosinophilic esophagitis knowledge measured on 8 true/false/I don't know questions where wrong or "I don't know" answers are given 0 points and correct answers are given 1 point. Minimum points=0 and Maximum points=8
Effectiveness (between-subjects) | Approximately 4 months
  Objective eosinophilic esophagitis knowledge measured on 8 true/false/I don't know questions where wrong or "I don't know" answers are given 0 points and correct answers are given 1 point. Minimum points=0 and Maximum points=8
Preparation for Decision Making (PrepDM) scale | Approximately 4 months
  Preparation for Decision making (PrepDM scale) score is a 10-item questionnaire and is scored on a 0-100 scale, where higher scores indicate participants being well prepared to make decisions after reviewing a decision aid (DA). The Prep-DM scale may be adapted slightly to meet the needs of the target population and the developed decision support tool.
Completion rates | Approximately 4 months
  Measured as the proportion of people that consented and completed all study measures, the pre-test, post-test, and 3-month follow-up survey

CONTACTS AND LOCATIONS:
Overall Officials: Joy Chang, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No